CLINICAL TRIAL: NCT04001140
Title: Enhancement of Emotion Regulation Skills in Vulnerable Adolescents at Risk for Addictions and Psychopathology Due to Risk Factors in the Family
Brief Title: Enhancement of Emotion Regulation Skills in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Christiana Theodorou, Principal Investigator, University of Cyprus
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: UCyprus
Record Dates: First submitted 2019-06-14; First posted 2019-06-27 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2019-06

CONDITIONS: Emotional Problem; Behavior Problem
Keywords: Emotion regulation; Prevention program; Adolescents; Physiological measurements; Internalizing problems; Externalizing problems
MeSH Terms: conditions — Mental Disorders; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The intervention group will take part in the sessions of the intervention, in which they learn different skills for the purpose of emotion regulation. All participants will complete the questionnaires and take part in the experiment again. This group prevention program, which is short-term, entailing 7 sessions, synthesizes techniques from three therapeutic models: Cognitive-Behavioral Therapy, Dialectical-Behavioral Therapy and Acceptance and Commitment Therapy.
  Interventions: Behavioral: Enhancement of emotion regulation skills
- Waiting-list group (No Intervention): The waiting-list group will receive the intervention 7 weeks after the intervention group finishes. The intervention group will finish the research in week 7, while the waiting-list group will start to attend the intervention. They will complete the questionnaires and the experiment.

INTERVENTIONS:
Behavioral: Enhancement of emotion regulation skills — Regarding the intervention, 7 sessions will be carried out. The main purpose is to help adolescents to enhance their emotion regulation, with the ultimate goal to decrease their risk of developing addictions and other psychopathology.
  Other Names: Cognitive-behavioral and dialectical-behavioral therapy
  Arms: Intervention group

SUMMARY:
For the current study, a prevention program is developed and applied to enhance the emotion regulation skills of adolescents. Before and after the application of the prevention program, all participants will be assessed for their emotion regulation ability via questionnaires and a physiological examination in which heart rate and skin conductance will be measured.

DETAILED DESCRIPTION:
The purpose of this research is to assess whether a short-term group intervention can enhance the emotion regulation skills of adolescents, when the family environment experiences stressful situations, psychopathology or substance abuse. This study aims to increase intervention effectiveness by examining effective approaches to train a crucial mechanism involved in emotional and behavior problems, which is emotion regulation. This research aims to develop a prevention program focused on the enhancement of adolescents' emotion regulation. Before and after the prevention program, participants will answer questionnaires and do a 5 minute psychophysiology experiment to evaluate their emotion regulation ability with both subjective and objective approaches. This prevention program, which is short-term, entailing 7 sessions, synthesizes techniques from three therapeutic models: Cognitive-Behavioral Therapy, Dialectical-Behavioral Therapy and Acceptance and Commitment Therapy. A short-term intervention was formulated and will be tested in the current study, with which is considered an advancement from previous similar interventions because of this synthesis and specific focus on emotion regulation skills, the lack of which can be considered a transdiagnostic risk factor across many psychological conditions and outcomes, including substance use. The main purpose is to help adolescents to enhance their emotion regulation, with the ultimate goal to decrease their risk of developing addictions and other psychopathology.

According to some classic theories of emotion, each emotion triggers a discrete pattern of behaviour, physiology, thoughts and feelings (Mauss & Robinson, 2009; Russell, 2003). This research will assess adolescents' emotion regulation through three dimensions: a) self-reported emotion reactivity (e.g. sensitivity, arousal/intensity and persistence), b) self-reported emotion regulation (e.g. self-blame, other-blame, rumination, catastrophizing, putting into perspective, positive refocusing, positive reappraisal, acceptance, planning, impulsivity, awareness and emotional clarity) and c) physiological (heart rate and skin conductance). These three dimensions will be assessed before and after the prevention program using relevant questionnaires and an experiment. The prevention program will focus on the enhancement of emotion regulation. However, it is expected that differences in the other two dimensions will also be found parallel to enhancement of emotion regulation skills.

Regarding the randomized control trial study, half of participants will take part in the intervention group and the other half in the waiting-list group. Participants will be divided into groups; each group of 5-10 adolescents (mixed male and female). Participants in the waiting-list group will receive the intervention when the intervention group finish the intervention. The questionnaires will be answered by all participants before and after the intervention and by those in the waiting list group. All participants will answer the questionnaires before and after a five week time interval during which the intervention will take place for the intervention group.

Physiological assessment of emotion processing will be of a 5 minutes duration, during an emotional imagery task, and participants participate twice -before and after the intervention for the intervention group, and two times with 5 weeks in between for the waiting-list group. The experiment will begin after a rest period which includes relaxation in the absence of any stimuli for 2 minutes (baseline) during which heart rate (HR) and skin conductance (SC) will be measured. Afterwards, participants will be asked to imagine six pre-standardized emotional scenarios, which three of them focusing on anger and three on fear situations, appropriate for their age. Participants will be given specific instructions on how to regulate their emotional responses to each scenario. Participants are given written instructions as to how they are to regulate elicited emotions during the different scenarios. Three different sets of emotion regulation instructions will be given to all participants: no guidance, acceptance and cognitive reappraisal. Participants will memorize each scenario prior to engaging in imagery and have to recall the scene as vividly as possible when each trial begins as prompted by the researcher. The duration of each imagery trial for each scenario is 30 seconds. Physiological measurements will be recorded during each scenario. More specifically, heart rate and skin conductance will be measured. Once this pre-intervention assessment is completed, the 7 sessions of group intervention will follow. In addition, at the end of each session participants will set a goal relevant to the skills which they have just learnt to practice at home as homework. For example, if the content of the session is the anger management, participants goal will be to start recognize their emotions and try to calm using different ways, and then when they are ready to express their emotions and try to find a functional solution.

ELIGIBILITY:
Inclusion criteria:

* Adolescents who have a family member with addiction problems (drug or alcohol use, gambling)
* Adolescents who have a family member with psychological problems (e.g. depression, anxiety disorder, bipolar disorder, etc.)
* Adolescents from stressful family environments (domestic violence, maltreatment, divorce, mourning, etc.)
* Participants are literate in Greek.

Exclusion criteria:

* Adolescents with severe addiction problems themselves (daily or weekly drugs use, such as cocaine, heroin, crystal meth, etc.)
* Adolescents with severe psychopathology (e.g. bipolar disorder, schizophrenia)
* Participants who are not literate in Greek.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Changes in difficulties of emotion regulation | Pre-Intervention (day 1), Post-Intervention (7 weeks after the pre-intervention), follow-up (6 months after the post-intervention)
  Self-reported measures for adolescents' emotion regulation skills: Difficulties in Emotion Regulation Scale (Gratz & Roemer, 2004). It is a brief, 36-item self-report questionnaire designed to assess multiple aspects of emotional dysregulation. Each item is rated on a 1 to 5 scale (1 =almost never and 4 = almost always). Higher scores suggest greater problems with emotion regulation. This questionnaire assesses six sub-scales: acceptance, goals, impulsivity, awareness, strategies and clarity.
Changes in enhancement of emotion regulation skills | Pre-Intervention (day 1), Post-Intervention (7 weeks after the pre-intervention), follow-up (6 months after the post-intervention)
  Self-reported measures for adolescents' emotion regulation: Cognitive Emotion Regulation Questionnaire (Garnefski, Kraaij, & Spinhoven, 2002). It is a 36-item questionnaire, consisting of 9 conceptually distinct subscales (Self-blame, Other-blame, Rumination, Catastrophizing, Putting into Perspective, Positive Refocusing, Positive Reappraisal, Acceptance and Planning). Each item is rated on a 1 to 5 scale (1 =almost never and 4 = almost always). Individual subscale scores are obtained by summing up the scores belonging to the particular subscale (ranging from 4 to 20). The higher the subscale score, the more a specific cognitive strategy is used.
Changes in heart rate | Pre-Intervention (day 1), Post-Intervention (7 weeks after the pre-intervention), follow-up (6 months after the post-intervention)
  Experiment: measured through heart rate
Psychophysiological changes in skin conductance | Pre-Intervention (day 1), Post-Intervention (7 weeks after the pre-intervention), follow-up (6 months after the post-intervention)
  Experiment: measured through skin conductance

SECONDARY OUTCOMES:
Depression symptoms | Pre-Intervention (day 1), Post-Intervention (7 weeks after the pre-intervention), follow-up (6 months after the post-intervention)
  Changes in the self-reported measure Youth Self-Report sub-scores of depression symptoms. This screening tool contains 13 questions to assess the depression symptoms, which are scored using a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). Higher scores suggest greater emotional problems.
Anxiety symptoms | Pre-Intervention (day 1), Post-Intervention (7 weeks after the pre-intervention), follow-up (6 months after the post-intervention)
  Changes in the self-reported measure Youth Self-Report sub-scores of anxiety symptoms. This screening tool contains 6 questions to assess the anxiety symptoms, which are scored using a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). Higher scores suggest greater anxiety problems.
Aggression problems | Pre-Intervention (day 1), Post-Intervention (7 weeks after the pre-intervention), follow-up (6 months after the post-intervention)
  Changes in the self-reported measure Youth Self-Report sub-scores of conduct disorder. This tool contains 15 questions to assess the conduct disorder, which are scored using a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). Higher scores suggest greater conduct problems.
Attention-Deficit/Hyperactivity Disorder symptoms | Pre-Intervention (day 1), Post-Intervention (7 weeks after the pre-intervention), follow-up (6 months after the post-intervention)
  Changes in the self-reported measure Youth Self-Report sub-scores of attention deficit/ hyperactivity disorder. This tool contains 7 questions to assess the attention deficit/ hyperactivity disorder, which are scored using a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). Higher scores suggest greater problems with attention deficit/ hyperactivity disorder.
Change in Nicotine Dependence | Pre-Intervention (day 1), Post-Intervention (7 weeks after the pre-intervention), follow-up (6 months after the post-intervention)
  Change in the Fagerstrom Test of Nicotine Dependence averaged scores. It contains six items that evaluate the quantity of cigarette consumption, the compulsion to use and dependence. Higher scores suggest nicotine dependence.
Change in alcohol consumption | Pre-Intervention (day 1), Post-Intervention (7 weeks after the pre-intervention), follow-up (6 months after the post-intervention)
  Change in the Alcohol Use Disorders Identification Test averaged scores

CONTACTS AND LOCATIONS:
Overall Officials: Christiana Theodorou, MSc., Principal Investigator — University of Cyprus; Georgia Panayiotou, Ph.D., Study Director — University of Cyprus
Locations (1):
- University of Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldin PR, Moodie CA, Gross JJ. Acceptance versus reappraisal: Behavioral, autonomic, and neural effects. Cogn Affect Behav Neurosci. 2019 Aug;19(4):927-944. doi: 10.3758/s13415-019-00690-7. PMID 30656602
- [Background] Milyavsky M, Webber D, Fernandez JR, Kruglanski AW, Goldenberg A, Suri G, Gross JJ. To reappraise or not to reappraise? Emotion regulation choice and cognitive energetics. Emotion. 2019 Sep;19(6):964-981. doi: 10.1037/emo0000498. Epub 2018 Sep 20. PMID 30234328
- [Background] Smith EN, Romero C, Donovan B, Herter R, Paunesku D, Cohen GL, Dweck CS, Gross JJ. Emotion theories and adolescent well-being: Results of an online intervention. Emotion. 2018 Sep;18(6):781-788. doi: 10.1037/emo0000379. Epub 2017 Dec 21. PMID 29265838
- [Background] Gross JJ. Emotion regulation: affective, cognitive, and social consequences. Psychophysiology. 2002 May;39(3):281-91. doi: 10.1017/s0048577201393198. PMID 12212647
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Sloan DM, Kring AM. Measuring changes in emotion during psychotherapy: conceptual and methodological issues. Clinical Psychology: Science and Practice 14: 307-322, 2007.
- [Background] Southam-Gerow MA. Emotion regulation in children and adolescents. New York: the Guilford Press, 2013.
- [Background] Gratz KL, Roemer L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment 26: 41-54, 2004.
- [Background] Thompson RJ, Dizen M, Berenbaum H. The Unique Relations between Emotional Awareness and Facets of Affective Instability. J Res Pers. 2009 Oct 1;43(5):875-879. doi: 10.1016/j.jrp.2009.07.006. PMID 20190861
- [Background] Feldman-Barrett L, Gross JJ, Christensen TC, Benvenuto M. Knowing what you're feeling and knowing what to do about it: mapping the relation between emotion differentiation and emotion regulation. Cognition and Emotion 15: 713-724, 2001.
- [Background] Marchesi C, Fonto S, Balista C, Cimmino C, Maggini C. Relationship between alexithymia and panic disorder: a longitudinal study to answer an open question. Psychother Psychosom. 2005;74(1):56-60. doi: 10.1159/000082028. PMID 15627858
- [Background] Leahy RL. A model of emotional schemas. Cognitive and Behavioral Practice 9: 177-190, 2002.
- [Background] Salovey P, Mayer JD, Goldman SL, Turvey C, Palfai TP. Emotional attention, clarity, and repair: exploring emotional intelligence using the trait meta-mood scale. In JW Pennebaker (Ed.), Emotion, disclosure, and health (pp. 125-154). Washington, DC: American Psychological Association, 1995.